CLINICAL TRIAL: NCT01901757
Title: An Open-label, Randomized, Single-dose, 2-way Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of HCP1201 Tablet in Healthy Volunteers
Brief Title: Single-dose, 2-way Crossover Open Study to Evaluate the Food Effect on the PK of HCP1201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MERO-102
Record Dates: First submitted 2013-07-07; First posted 2013-07-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP1201, Fasted followed by fed (Experimental): HCP1201 dosing in the fasted state followed by fed dosing
  Interventions: Drug: HCP1201, Fasted followed by fed; Drug: HCP1201, Fed followed by fasted
- HCP1201, Fed followed by fasted (Experimental): HCP1201 dosing in the fed state followed by fasted dosing
  Interventions: Drug: HCP1201, Fasted followed by fed; Drug: HCP1201, Fed followed by fasted

INTERVENTIONS:
Drug: HCP1201, Fasted followed by fed — There are 2 administration periods with 7 days of wash-out. In period 1, the subjects will receive a single oral dose of HCP1201 under fasted condition. In period 2, the subjects will receive a single oral dose of HCP1201 under fed condition.
Drug: HCP1201, Fed followed by fasted — There are 2 administration periods with 7 days of wash-out. In period 1, the subjects will receive a single oral dose of HCP1201 under fed condition. In period 2, the subjects will receive a single oral dose of HCP1201 under fasted condition.

SUMMARY:
To investigate the effect of food in healthy male volunteers who receive HCP1201 tablet in fed versus fasted condition

DETAILED DESCRIPTION:
An open-label, randomized, single-dose crossover study to evaluate the effect of food on the pharmacokinetics of HCP1201 tablet in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 20~55 years
2. The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
3. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
4. Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Glomerular filtration rate is under 60ml/min which is calculated by serum creatinine value.
3. Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.
4. Systolic Blood Pressure: lower than 90mmHg or higher than 150mmHg, Diastolic Blood Pressure: lower than 60mmHg or higher than 100mmHg
5. History of relevant drug allergies or clinically significant hypersensitivity reaction.
6. History of drug abuse or positive drug screening.
7. Participation in other drug studies within 60days prior to the drug administration.
8. Whole blood donation within 60 days, blood component donation within 30 days or who got transfusion within 30days.
9. Subjects who took prescription drugs within 14 days from the patient screening or non-prescription medicine within 7 days which can affect the result of this clinical trial (acceptable according to the investigator's judgement)
10. Subjects who took medicines(e.g. proton pump inhibitor, rifampicin, oriental medicines, etc.) within 30days that can affect absorption, distribution, metabolism, elimination of metformin/rosuvastatin.
11. Intake of more than 140g of alcohol per week or who can't abstain from alcohol during the trial.
12. Subjects who smoke more than 10 cigarettes per day or who can't quit smoking during the trial.
13. Positive screening on Hepatitis B surface antigen(HBsAg), anti-Hepatitis C virus(HCV) or anti-Human immunodeficiency virus(HIV).
14. Genetic myopathic disorder or related family history, medical history of myopathic disorder caused by medication.
15. Clinically inappropriate laboratory test result.
16. Clinically inappropriate electrocardiogram result.
17. Subjects who judged ineligible by the investigator.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Metformin, rosuvastatin Cmax, AUClast | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

SECONDARY OUTCOMES:
Metformin, rosuvastatin Tmax | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin T1/2 | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin AUCinf | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin CL/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h
Metformin, rosuvastatin Vd/F | pre-dose, post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ryul Kim, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea